CLINICAL TRIAL: NCT02704312
Title: A Feasibility Study of Patient Comfort and Dosimetry Evaluation in Prone Breast Radiotherapy.
Brief Title: Dosimetric Comparison of Doses in Both Positions (Prone and Decubitus) for Patient With Breast Cancer
Acronym: PROCUBITUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Start of the Principal Investigatoir
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15/ B/ 25
Record Dates: First submitted 2016-03-01; First posted 2016-03-10 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy techniques (Experimental): Quantitative Physics: dosimetric comparison of doses in target volumes and organs at risk. The technique used is that of which the dose on the organs at risk is as low as possible, and whose dose to the target volume is the closest possible to the prescribed dose (100% of the prescribed dose)
  Interventions: Radiation: Radiotherapy by Prone and decubitus

INTERVENTIONS:
Radiation: Radiotherapy by Prone and decubitus — Dosimetric comparison of doses in target volumes and organs at risk

SUMMARY:
Compare dosimeters in both positions (prone and decubitus) for each patient

DETAILED DESCRIPTION:
Quantitative Physics: dosimetric comparison of doses in target volumes and organs at risk. The technique used is that of which the dose on the organs at risk is as low as possible, and whose dose to the target volume is the closest possible to the prescribed dose (100% of the prescribed dose).

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary breast cancer and in whom conservative post- surgery radiation therapy for breast cancer is prescribed.
* Patients aged over 18 years
* Patients with indication for conservative surgery.
* Resection should be in healthy margin.
* Women of childbearing potential must satisfy a negative pregnancy test at the screening visit and use effective contraception as determined by the physician of the patient throughout the study.

Exclusion Criteria:

* Minor Patient
* Patients whose tumor resection is incomplete
* Patients with an indication of mastectomy
* Patients with a history of radiation therapy of the chest
* Pregnant women, lactating, or of childbearing age without effective contraception.
* Patients who had more than 4 scanners in one year. ( Scanner cervical , thoracic, or abdominal
* Patients with an incompatible condition with monitoring protocol (psychiatric disorder, uncontrolled disease).
* Patient unable to respond to a questionnaire

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Quantitative Physics: dosimetric comparison of doses in target volumes and organs at risk | From baseline to 5 weeks

SECONDARY OUTCOMES:
Quality of Life Questionnaire | Baseline and Follow up month 3, 12, 24 and 36

CONTACTS AND LOCATIONS:
Overall Officials: Vincent VINH HUNG, MD, Principal Investigator — CHU de Martinique
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No